CLINICAL TRIAL: NCT01839162
Title: RAdiation Dose In percutAneuos Coronary Procedures Through TransradIal apprOach Using Dedicated radiatioN Shields (The RADIATION Study)
Brief Title: RAdiation Dose In percutAneuos Coronary Procedures Through TransradIal apprOach Using Dedicated radiatioN Shields
Acronym: RADIATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Alessandro Sciahbasi, MD, Interventional Cardiologist, Ospedale Sandro Pertini, Roma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASLRMB-Pertini1
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Myocardial Ischemia
Keywords: Transradial approach; shield drape; radiation; PTCA
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pelvic drape (Experimental): Pelvic shield drape over the patient
  Interventions: Procedure: Coronary angiography; Procedure: PCI; Procedure: Right approach; Procedure: Left approach
- Arm drape (Experimental): Right radial arm drape over the patient
  Interventions: Procedure: Coronary angiography; Procedure: PCI; Procedure: Right approach; Procedure: Left approach
- Pelvic and arm drape (Experimental): Pelvic and arm drpaes placed over the patient
  Interventions: Procedure: Coronary angiography; Procedure: PCI; Procedure: Right approach; Procedure: Left approach
- No drapes (Sham Comparator): Standard radioprotection devices
  Interventions: Procedure: Coronary angiography; Procedure: PCI; Procedure: Right approach; Procedure: Left approach

INTERVENTIONS:
Procedure: Coronary angiography — Diagnostic coronary angiography
Procedure: PCI — Percutaneous coronary intervention
Procedure: Right approach — Right transradial access
Procedure: Left approach — Left transradial access

SUMMARY:
During percutaneous coronary interventions standard operator radio-protection is generally ensured using a lead apron, a thyroid lead collar, low leaded flaps, an upper mobile leaded glass suspended from the ceiling and leaded glasses. Previous studies showed that adding a bismuth-barium radiation shield drape on the patient right arm or using a pelvic lead shield on the patient, the radiation dose adsorbed by operators was significantly reduced even if was higher compared to transfemoral approach. No studies evaluated the effect of both adjunctive shields placed in the same patient.

Aim of our randomized study is to evaluate if the combination of a shield drape on the patient right arm and a pelvic lead shield during transradial percutaneous coronary procedures may reduce the radiation dose adsorbed by operators compared to the use of only one shield or none.

All patients who underwent to percutaneous coronary diagnostic or interventional procedures will be enrolled in this randomized study. Eligible patients will be randomized (using a computer generated randomization sequence) in 4 groups:

1. use of a pelvic shield drape
2. use of a shield drape on the patient right arm
3. use of a pelvic shield drape and a shield drape on the patient right arm
4. Any adjunctive shield drape (only standard radio-protection) For each group a further internal randomization will be performed in order to compare the right or left radial transradial approach.

Each operator will be equipped with dedicated dosimeters placed at left wrist and at thorax level outside the lead apron. Since December 2013 the operators are equipped with a further dosimeter at head level.

Primary end-point of the study is the radiation dose adsorbed at wrist and thorax by operators and detected by the electronic dosimeters.

Secondary end-point are:

1. Radiation dose adsorbed by operators according to the radial access (right versus left)
2. Radiation dose adsorbed by the patients
3. Radiation dose adsorbed at head level.

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent to percutaneous coronary diagnostic or interventional procedures will be enrolled in this randomized study

Exclusion Criteria:

1. Previous coronary artery by-pass
2. Acute ST elevation myocardial infarction
3. Hemodynamic instability or cardiogenic shock
4. Ischemic Allen test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Radiation dose adsorbed by operators | During procedure
  Primary end-point of the study is the radiation dose adsorbed at wrist and thorax by operators and detected by the electronic dosimeters

SECONDARY OUTCOMES:
Radiation dose adsorbed by operators according to the radial access (right versus left) | During procedure
  Radiation dose adsorbed by operators according to the radial access (right versus left)
Radiation dose adsorbed by the patients | During procedure
  Radiation dose adsorbed by the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Sandro Pertini - ASL RMB- UOSD Emodinamica, Rome, Rome, Italy